CLINICAL TRIAL: NCT05706272
Title: Secure And Focused Primary Care for Older pEople (SAFE) - A Proactive Trial
Brief Title: Secure and Focused Primary Care for Older pEople
Acronym: SAFE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other); Region Jönköping County (Other Government)
Responsible Party: Principal Investigator, Anna Segernas, PhD MD, Linkoeping University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-03388-01
Record Dates: First submitted 2023-01-09; First posted 2023-01-31 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Frailty
Keywords: Frailty; Primary care; Geriatrics; Comprehensive geriatric assessment
MeSH Terms: conditions — Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Intervention Model Description: The study will include 26 intervention primary care practices and 25 matched control practices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention primary care practices (Experimental): The participants in the intervention primary care practices arm will receive a holistic CGA using the PASTEL assessment tool. An "elderly team" including a doctor and nurse will work around the patient. The intervention includes increased care coordination.
  Interventions: Other: Comprehensive geriatric assessment (CGA)
- Matched control primary care practices (Active Comparator): The participants in the matched control primary care practices arm will receive care as usual at the matched control primary care centers.
  Interventions: Other: Care as usual

INTERVENTIONS:
Other: Comprehensive geriatric assessment (CGA) — The intervention includes a holistic comprehensive geriatric assessment using the PASTEL assessment tool that includes medical, psychiatric, functional and social aspects. Physical tests will include function, risk of falling, hand muscle strength, Timed up and Go (TUG), chair-stand test, blood pressure, saturation and BMI. A proactive person centered care plan will be established based on identified needs and the patients own priorities. A nurse will coordinate the care in the elderly team at the intervention practice with access to rehabilitation staff such as physiotherapist and occupational therapist. Follow-ups at the primary care practices will be carried out in accordance with the study plan. To strengthen care coordination, contact will be taken with other health care providers before the follow-ups.
  Arms: Intervention primary care practices
Other: Care as usual — The control group will receive care as usual at the matched control primary care centers
  Arms: Matched control primary care practices

SUMMARY:
The population worldwide is aging. The demographic change is challenging to health care organizations and highlights the need for effective preventive and proactive care models in primary care, especially for older people. This study, "Secure and focused primary care for older people" (SAFE), investigates the effectiveness of a new proactive care model based on comprehensive geriatric assessment (CGA) in primary care in a population with high risk of hospitalisation.

DETAILED DESCRIPTION:
Background and Aim

The number of old people is rising and in Sweden, approximately 20% of the population is older than 65 years. In 2050, the number of people 85 years and above, is expected to have doubled [1]. The demographic change is challenging to future healthcare systems [2]. The prevailing strategy for reducing the healthcare impact of an ageing population has been 'compression of morbidity', to extend the healthy period of life, and delay disability until a brief period at the end of life [3]. Thus, preventative and proactive primary care is central in meeting future challenges such as an aging population and highlights the need for effective preventive and proactive care models in primary care, especially for older people. This study, "Secure and focused primary care for older people" (SAFE), investigates the effectiveness of a new proactive care model in primary care in a population with high risk of hospitalisation.

Comprehensive geriatric assessment (CGA) is considered gold standard in evaluation and caring for old in-hospital patients [4]. CGA is described as a multidimensional, multidisciplinary and holistic evaluation of the health status of an older person, together with the formation of a care plan based on individual needs and preferences [4]. Data from outpatients in geriatric care has shown that CGA may delay the progression of frailty, but the study population was quite small [5].There is evidence that CGA can decrease the need of inpatient care and nursing home admissions. Some studies suggest that comprehensive care programs can be cost-effective. They also seem to be widely accepted and increase patient satisfaction [6,7]. However, results are conflicting and meta-analyses suffer from the lack of a universal definition of frailty and the great variation of interventions, outcome measures and scales to measure frailty. Still, both NICE guidelines and the ICOPE recommendations of the WHO include CGA for older people with frailty and/or multimorbidity [8].

In a previous study, "Proactive healthcare for frail elderly persons", a predictive statistical model that identified individuals, 75 years and above, with high risk for hospitalisation during the coming 12 months, was validated [9]. The effectiveness of CGA adapted to primary care using the new CGA tool: the Primary care Assessment Tool for Elderly (PASTEL), delivered to older adults with identified high risk for hospitalisation, was evaluated [10]. This pragmatic multicenter trial comprised nine intervention practices and ten matched control practices in the county council of Östergötland, Sweden, in 2017-2019. No specific intervention measures beyond the CGA assessment with PASTEL were described or analyzed in the study. Follow-up was part of ordinary clinical routine. Which specific interventions in primary care that really make a difference to reduce risk for hospitalisation and improve quality of life for old outpatients remains to be explored.

The main aim of the present study is to examine whether a proactive care model with comprehensive geriatric assessment (CGA) in primary care with additional long-term care coordination and increased patient participation, contributes to reduced inpatient care and/or increased quality of life among community-dwelling older people. The CGA used in this study will be based on the instrument "the Primary Care Assessment Tool for Elderly" (PASTEL).

Design and Method

This is a prospective, multi-center trial that will be carried out in two regions in Sweden (Östergötland and Jönköping). The study will include 26 intervention primary care practices and 25 matched control primary care practices. Data will be collected at baseline, at one year follow-up (12 months) and at two year follow-up (24 months).

Participants will be identified through a statistical prediction model based on age, health care use and diagnostics data covering the previous year. A risk score for future morbidity and health care need will be calculated and the participants with the highest risk scores (top 15%) will be invited to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* 75 years or older
* community dwelling (living in own home)
* Top 15% of risk score calculation

Exclusion Criteria:

- Persons living in nursing homes

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of in-hospital days | 24 months
  Total number of days that a patient is admitted to hospital

SECONDARY OUTCOMES:
Number of in-hospital episodes | 24 months
  Number of times that a patient is admitted to hospital (regardless of length of stay)
Number of health care visits | 24 months
  Number of visits that a patient makes to a health care provider (hospital and primary care)
Number of persons living in nursing homes | 24 months
  Number of persons living in a nursing home
Time to event (when moving to nursing home) | 24 months
  The time when a person needs to move from own home to a nursing home
Mortality | 24 months
  All cause mortality
Health care costs | 24 months
  Total health care costs including hospital care and primary care
Health related quality of life (HRQoL) | 24 months
  HRQoL collected through the EQ-5D-5L
Cost-effectiveness, cost/QALY | 24 months
  Health economic calculation of the cost-effectiveness of the intervention including both health care costs and HRQoL data
Sense of safety and control | 24 months
  The patients sense of safety and control will be collected using the ASCOT instrument
Health related quality of life (HRQoL) | 24 months
  HRQoL collected through the RAND-36

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Region Jönköping, Jönköping
  - Region Östergötland, Linköping

IPD SHARING:
Plan to Share IPD: Undecided
Data may be made available upon request when the study is completed following the laws for sharing patient data.

REFERENCES:
- [Background] Socialstyrelsen, Vård om omsorg om äldre, 2020. https://www.socialstyrelsen.se/globalassets/sharepoint-dokument/artikelkatalog/ovrigt/2020-3-6603.pdf.
- [Background] Partridge L, Deelen J, Slagboom PE. Facing up to the global challenges of ageing. Nature. 2018 Sep;561(7721):45-56. doi: 10.1038/s41586-018-0457-8. Epub 2018 Sep 5. PMID 30185958
- [Background] Seals DR, Justice JN, LaRocca TJ. Physiological geroscience: targeting function to increase healthspan and achieve optimal longevity. J Physiol. 2016 Apr 15;594(8):2001-24. doi: 10.1113/jphysiol.2014.282665. Epub 2015 Mar 11. PMID 25639909
- [Background] Parker SG, McCue P, Phelps K, McCleod A, Arora S, Nockels K, Kennedy S, Roberts H, Conroy S. What is Comprehensive Geriatric Assessment (CGA)? An umbrella review. Age Ageing. 2018 Jan 1;47(1):149-155. doi: 10.1093/ageing/afx166. PMID 29206906
- [Background] Mazya AL, Garvin P, Ekdahl AW. Outpatient comprehensive geriatric assessment: effects on frailty and mortality in old people with multimorbidity and high health care utilization. Aging Clin Exp Res. 2019 Apr;31(4):519-525. doi: 10.1007/s40520-018-1004-z. Epub 2018 Jul 23. PMID 30039453
- [Background] Hopman P, de Bruin SR, Forjaz MJ, Rodriguez-Blazquez C, Tonnara G, Lemmens LC, Onder G, Baan CA, Rijken M. Effectiveness of comprehensive care programs for patients with multiple chronic conditions or frailty: A systematic literature review. Health Policy. 2016 Jul;120(7):818-32. doi: 10.1016/j.healthpol.2016.04.002. Epub 2016 Apr 11. PMID 27114104
- [Background] Pilotto A, Cella A, Pilotto A, Daragjati J, Veronese N, Musacchio C, Mello AM, Logroscino G, Padovani A, Prete C, Panza F. Three Decades of Comprehensive Geriatric Assessment: Evidence Coming From Different Healthcare Settings and Specific Clinical Conditions. J Am Med Dir Assoc. 2017 Feb 1;18(2):192.e1-192.e11. doi: 10.1016/j.jamda.2016.11.004. Epub 2016 Dec 31. PMID 28049616
- [Background] National Guideline Centre (UK). Multimorbidity: Assessment, Prioritisation and Management of Care for People with Commonly Occurring Multimorbidity. London: National Institute for Health and Care Excellence (NICE); 2016 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK385543/ PMID 27683922
- [Background] Marcusson J, Nord M, Dong HJ, Lyth J. Clinically useful prediction of hospital admissions in an older population. BMC Geriatr. 2020 Mar 6;20(1):95. doi: 10.1186/s12877-020-1475-6. PMID 32143637
- [Background] Nord M, Lyth J, Alwin J, Marcusson J. Costs and effects of comprehensive geriatric assessment in primary care for older adults with high risk for hospitalisation. BMC Geriatr. 2021 Apr 21;21(1):263. doi: 10.1186/s12877-021-02166-1. PMID 33882862